CLINICAL TRIAL: NCT04227977
Title: Volume Optimization Incorporating Negative Pressure Diuresis in Heart Failure (VOID-HF)
Acronym: VOID-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 3ive Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VOID-HF
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Cardiorenal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): JuxtaFlow
  Interventions: Device: JuxtaFlow System

INTERVENTIONS:
Device: JuxtaFlow System — The JuxtaFlow System consists of proprietary ureteral catheters deployed endoscopically over the wire to deliver mild controlled negative pressure into the renal pelvis.

SUMMARY:
The Cardiorenal Syndrome during Acute decompensated heart failure (ADHF) with persistent congestion despite high dose IV diuretic therapy is associated with remarkable morbidity, which can include the need for renal dialysis or ultrafiltration, an increased length of stay, and high mortality rates. The aims and purpose of this feasibility clinical research trial are: 1. to evaluate the safety profiles associated with performing negative pressure diuresis for the treatment of hypervolemia associated with the cardiorenal syndrome during ADHF with persistent congestion despite high dose IV diuretic therapy via the investigational JuxtaFlow® System, and 2. to evaluate the effectiveness of the investigational JuxtaFlow System in treatment of hypervolemia associated with ADHF.

DETAILED DESCRIPTION:
The Cardiorenal Syndrome during Acute decompensated heart failure (ADHF) with persistent congestion despite high dose IV diuretic therapy is associated with remarkable morbidity, which can include the need for renal dialysis or ultrafiltration, an increased length of stay, and high mortality rates. The primary renal adjuvant therapies for presistent congestion despite high dose IV diuretic therapy are ultrafiltration and dialysis. Unfortunately, clinical decongestion is uncommon in this population despite aggressive therapies. Negative pressure diuresis in the renal pelvis has the potential to treat hypervolemia associated with ADHF by increasing renal filtration and increased urine output.

Primary endpoint: The characterization of the type, frequency, severity, and device-relatedness of adverse events (AEs) associated with the placement, use, and removal of the JuxtaFlow System and a 28-day post-treatment actuarial follow up.

Secondary endpoints: a) Increase in urine output from baseline to discontinuation of treatment with the JuxtaFlow System. b) Reduction of congestion (as measured by change in BNP) during the course of the treatment with the JuxtaFlow System. c) The relative change in creatinine clearance from baseline to treatment period after 24 hours of treatment or until discontinuation of the investigational treatment using each study subject as their own control. The change in creatinine clearance from the baseline period to the 24 hour post End of Treatment (EOT) period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥22 years of age
2. Patients admitted with primary diagnosis of ADHF
3. Persistent volume overload with venous congestion despite at least 24 hours of IV diuretic therapy, including either a single bolus ≥ 100 mg or continuous drip ≥ 10 mg/hour of furosemide equivalent, where:

   1. Volume overload defined by the presence of pulmonary edema, 2+ peripheral edema, or orthopnea
   2. Venous congestion defined by at least one of the following:

   i. Jugular venous pressure > 10 cm on physical exam ii. Central venous pressure > 10 mmHg iii. Pulmonary capillary wedge pressure > 22 mmHg c) Evidence of low natriuretic response to high dose diuretic therapy defined by spot urine sodium < 70 mmol
4. Ability to have the JuxtaFlow® System catheters placed at bedside
5. Anticipated to have an inpatient hospital admission that is ≥ 72 hours
6. Patients that are willing and able to provide informed consent for this research trial, or if the patient is not able to provide consent due to their clinical condition, a legal guardian, spouse, or next of kin to the patient with medical power of attorney that is willing to provide consent for the patient's participation in this research trial
7. Patients who agree to comply with the study procedures and specified evaluations

Exclusion Criteria:

1. Females who are pregnant or nursing mothers
2. Creatinine > 3.0 mg/dL at admission to the hospital
3. Systolic blood pressure < 100 mmHg at the time of enrollment
4. Clinical instability likely to require the addition of intravenous vasoactive drugs, vasodilators and/or inotropic agents.
5. Alternative explanation for the renal impairment causing the persistent volume overload, such as obstructive nephropathy, contrast induced nephropathy, or acute tubular necrosis
6. Any patient with an eGFR < 15 ml/min or prior diagnosis of CKD 5
7. Any patient presenting with hematuria as defined by urine dipstick reading of > 1+ blood
8. Any patient presenting with proteinuria as defined by urine dipstick reading of > 3+ protein.
9. Any patient that would not potentially benefit from this therapy in the opinion of the investigator
10. Any patient with a current upper or lower urinary tract infection (tested during pre-screening)
11. Any patient with a malignancy of the upper urinary tract
12. Any patient who are currently experiencing unexplained/unexpected proteinuria as determined by the investigator
13. Any patient with a current unrepaired ureteral avulsion as determined by the investigator
14. Any patient that would require an MRI between enrollment and completion of the post-treatment baseline period
15. Any secondary condition as determined by the investigator that would place the subject at an increased risk, or preclude the subject's full compliance with the study procedures, including injuries to the urinary organs and/or external genitals
16. Any use of an iodinated radiocontrast material in the past 72 hours prior to study enrollment or anticipated use of intravenous contrast during the current hospitalization.
17. Pre-enrollment ultrasound revealing any of the following:

    1. Congenital abnormality in either kidney
    2. Only one kidney
    3. Presence of debris, stones or an obstruction in the renal pelvis, ureter or urinary tract
18. Current or planned treatment with an investigational drug (IND), device (IDE), or other investigational intervention within 3 months prior to or during participation in this clinical trial

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Device related adverse events | 28 days
  The characterization of the type, frequency, severity, and device-relatedness of adverse events (AEs) associated with the placement, use, and removal of the JuxtaFlow System and a 28-day post-treatment follow up.

SECONDARY OUTCOMES:
Urine output | 24 hours
  The change in urine output from baseline to discontinuation
Congestion | 24 hours
  The change in congestion (as measured by change in BNP) during the course of treatment
Creatinine Clearance | 24 hours
  The change in creatinine clearance from baseline to discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Tang, MD, Principal Investigator — The Cleveland Clinic; Alex Parker, MD, Principal Investigator — Univ. of Florida, Gainesville; Wayne Old, MD, Principal Investigator — Sentara Norfolk General Hospital; Shweta Bansal, MD, Principal Investigator — Univ. of Texas Health, San Antonio
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Cleveland Clinic, Cleveland, Ohio
  - Univ. of Texas Health, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No